CLINICAL TRIAL: NCT01656603
Title: A Multicenter Safety Study of Unlicensed, Investigational Cryopreserved Cord Blood Units Manufactured by the National Cord Blood Program and Provided for Unrelated Hematopoietic Stem Cell Transplantation of Pediatric and Adult Patients
Brief Title: Safety Study of Unlicensed IND Cord Blood Units Manufactured by the National Cord Blood Program for Unrelated Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Blood Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6637-01; NCT01861093 (obsolete NCT alias)
Record Dates: First submitted 2012-07-31; First posted 2012-08-03 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-03

CONDITIONS: Infusion Reactions
Keywords: cord blood; transplantation; stem cells; adverse event

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- unlicensed CBU (Experimental): The Principal Investigators will be the transplant physicians at participating US transplant centers
  Interventions: Biological: unlicensed CBU

INTERVENTIONS:
Biological: unlicensed CBU — infusion of unlicensed cord blood units

SUMMARY:
This study will evaluate the safety of infusion of the investigational cord blood units by carefully documenting all infusion-related problems.

DETAILED DESCRIPTION:
The primary aim of this study is to examine the safety of administration of the unlicensed investigational NCBP hematopoietic progenitor cell-cord blood (HPC-CORD BLOOD) products in a multi-institution setting. Therefore, the study will evaluate prospectively the incidence of serious adverse reactions as well as the incidence of all infusion related reactions after administration of the unlicensed, investigational NCBP CBU.

Definitions of Infusion-related adverse reactions:

Mild - Moderate: reactions during or after the infusion of the cord blood (CB) product that require some medical intervention but do not affect the overall patient status or outcome.

Severe: serious, life-threatening or fatal infusion reactions, requiring major medical intervention. These include: anaphylactic shock, acute cardiac, pulmonary or renal failure, seizures, patient transfer to the Intensive Care Unit, or death within 48 hours of the CB infusion. Adverse Reactions will also be classified by grade, according to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Patients with disorders affecting the hematopoietic system that are inherited, acquired, or result from myeloablative treatment.
2. Patients: Patients of any age and either gender
3. Cord blood product manufactured by the NCBP (at least one, if the graft contains more than one units)

Exclusion Criteria:

1. Patients who are receiving licensed cord blood products (only)
2. Patients who are receiving unlicensed cord blood products from other banks (only)
3. Patients who are transplanted at non-US transplant centers
4. Patients who are receiving cord blood products that will be "manipulated" post-thaw (e.g., ex vivo expansion, incubation in vitro, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9999 (Estimated)
Dates: Start 2012-02; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of infusion-related reactions | within 48 hours of infusion
  The primary aim of this study is to examine the safety of administration of the unlicensed investigational cord blood products in a multi-institution setting. The study will evaluate prospectively the incidence of serious adverse reactions as well as the incidence of all infusion related reactions after administration of the unlicensed, investigational NCBP cord blood units.

SECONDARY OUTCOMES:
engraftment | six months after transplant
  This outcome will evaluate engraftment of unlicensed cord blood units

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Shi, MD, Principal Investigator — NY Blood Center
Locations (71):
- United States (71):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA Healthcare, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Stanford Health Care, Stanford, California
  - The Children's Hospital of Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Presbyterian / St. Luke's Medical Center, Denver, Colorado
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemour's Children's Clinic and Hospital, Jacksonville, Florida
  - University of Miami Health System Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - Florida Hospital, Florida Center for Cellular Therapy, Orlando, Florida
  - All Children's Hospital, John Hopkins Medicine, St. Petersburg, Florida
  - Northside Hosptal, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Indiana University, Indianapolis, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - National Institutes of Health, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Instistute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Barnes-Jewish Hospital at University of Washington / Sireman Cancer Center, St Louis, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - Northwell Health - North Shore University Hospital, Lake Success, New York
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - New York Presbyterian Hospital WCMC, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Arthur G. James Cancer Hospital, Columbus, Ohio
  - Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Southwestern Regional Medical Center, Tulsa, Oklahoma
  - Doernbecher Children's Hospital / Oregon Health & Science University, Portland, Oregon
  - Penn State Health / Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hopsital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St Jude Children's Research Center, Memphis, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - Methodist Hospital / Texas Transplant Institute, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center / Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No